CLINICAL TRIAL: NCT00856791
Title: Phase II Single-arm Study of ON 01910.Na by 2-hr Infusion in Patients With Recurring Platinum-resistant Ovarian Cancer
Brief Title: Effect of 2-h Infusion of ON 01910.Na in Ovarian Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Traws Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Onconova 04-12
Record Dates: First submitted 2009-03-04; First posted 2009-03-06 (Estimated); Results first posted 2013-01-08 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-06

CONDITIONS: Ovarian Cancer
Keywords: Ovarian; Cancer; Cisplatin; Carboplatin
MeSH Terms: conditions — Ovarian Neoplasms; Neoplasms | interventions — ON 01910

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ON 01910.Na (Experimental): 3200 mg ON 01910.Na administered intravenously over 2 hours on days 1, 4, 8, 11, 15, and 18 of 28-day cycle
  Interventions: Drug: ON 01910.Na

INTERVENTIONS:
Drug: ON 01910.Na
  Other Names: rigosertib; rigosertib sodium

SUMMARY:
ON 01910.Na has undergone preclinical and clinical phase I studies showing activity in patients with progressing ovarian cancer resistant to platinum-based chemotherapies. This study will look at a larger population of patients to determine whether treatment with ON 01910.Na has an effect on progression free survival rates in patients with platinum-resistant ovarian cancer. ON 01910.Na will be given as an intravenous infusion over 2 hours on days 1, 4, 8, 11, 15, and 18 of a 28-day cycle. Patients will be treated for 6 or more cycles.

DETAILED DESCRIPTION:
This is a Phase II single arm study of ON 01910.Na to be administered as a 2-hour infusion biweekly to patients with progressive ovarian cancer resistant to platinum-based therapy.

The primary objective is to evaluate progression-free survival (PFS). The secondary objectives are to document other measures of outcome [objective response rate (ORR), duration of response, duration of stable disease, and overall survival (OS)], and tolerability of study drug.

Thirty-seven (37) patients with progressive ovarian cancer resistant to platinum-based therapy will be enrolled in a single arm study and treated with ON 01910.Na administered as a 2-hour infusion on Days 1, 4, 8, 11, 15 and 18 of a 28-day cycle. Patients will be treated until disease progression or withdrawal for other causes (unacceptable toxicity, patient or investigator decision) with ON 01910.Na. Toxicity will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE v3.0). Progression-free survival, objective response, duration of response, and duration of stable disease will be assessed using RECIST (Response Evaluation Criteria in Solid Tumor) guidelines, as well as overall survival. Grades 3 and 4 hematologic toxicities, grade >2 non-hematologic toxicities will be monitored. A futility analysis will be performed after 17 evaluable patients are enrolled and evaluated for overall objective response. If 3 or fewer objective response (CR and PR) are observed, the study will be closed to further accrual and deemed futile. An extension study for an additional 25 weeks with complete monitoring will be considered for patients who have not progressed by week 25.

The ON 01910.Na dose to be used in this study (2-hour infusions of 2400 or 3200 mg twice weekly for 3 weeks of a 4-week cycle) was selected based on the maximum tolerated doses and activities documented in phase 1 protocols.

ELIGIBILITY:
Inclusion Criteria:

* Women with ovarian cancer at least 18 years old with measurable disease who have shown recurrent disease within 6 months of the last dose of cisplatin- or carboplatin-based chemotherapy. Measurable disease will be defined as lesions that can be accurately measured in at least one dimension with longest diameter ≥ 20 mm using conventional techniques or ≥ 10 mm with spiral CT scan.
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0, 1 or 2.
* No more than 3 prior chemotherapy regimens.
* Disease-free period of more than 5 years from prior malignancies other than ovarian (except curatively treated basal cell carcinoma, squamous cell carcinoma of the skin,or carcinoma in situ of the cervix).
* All female patients of childbearing potential must use at least one form of contraception as approved by the Investigator prior to study entry and for up to 30 days beyond the last administration of study drug.
* Women of childbearing potential must have a negative serum βHCG pregnancy test at screening.
* Willing to adhere to the prohibitions and restrictions specified in this protocol.
* Patient (or her legally authorized representative) must have signed an informed consent document.

Exclusion Criteria:

* Evidence of complete or partial bowel obstruction.
* Need for IV hydration or Total Parenteral Nutrition.
* Inability to comply with study and/or follow-up procedures.
* Life expectancy of less than 12 weeks.
* Prior radiotherapy to greater than one third of hematopoietic sites.
* Uncontrolled intercurrent illness including, but not limited to symptomatic congestive heart failure, unstable angina pectoris or cardiac arrhythmia.
* Active infection not adequately responding to appropriate therapy.
* Hyponatremia (defined as serum sodium value of <134 mEq/L).
* Total bilirubin ≥ 1.5 mg/dL not related to hemolysis or Gilbert's disease, AST/ALT or alkaline phosphatase ≥ 2 X ULN.
* Serum creatinine ≥ 2.0 mg/dL.
* ANC < 1500/mm3, platelets < 100,000/mm3; hemoglobin less than 9 g/dL.
* Ascites requiring active medical management including paracentesis for more than twice a month.
* Women patients who are pregnant or lactating or have a positive serum βHCG pregnancy test at screening.
* Major surgery without full recovery or major surgery within 3 weeks of ON 01910.Na treatment start.
* Uncontrolled hypertension (defined as a systolic pressure ≥ 160 and/or a diastolic pressure ≥ 110).
* New onset seizures (within 3 months prior to the first dose of ON 01910.Na) or poorly controlled seizures.
* Brain metastases including any of the following:

  1. Evidence of cerebral edema by CT scan or MRI.
  2. Evidence of disease progression on prior imaging studies.
  3. Requirement for steroids.
  4. Clinical symptoms of brain metastases.
* Any concurrent and/or within 4 weeks of the first dose of study drug investigational agent or chemotherapy, radiotherapy or immunotherapy.
* Psychiatric illness/social situations that would limit the patient's ability to tolerate and/or comply with study requirements.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2009-03; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory P. Sutton, MD, Principal Investigator — St. Vincent Gynecologic Oncology, Indianapolis, IN
Locations (1):
- St. Vincent Gynecologic Oncology, Indianapolis, Indiana, United States

REFERENCES:
- [Background] Jimeno A, Li J, Messersmith WA, Laheru D, Rudek MA, Maniar M, Hidalgo M, Baker SD, Donehower RC. Phase I study of ON 01910.Na, a novel modulator of the Polo-like kinase 1 pathway, in adult patients with solid tumors. J Clin Oncol. 2008 Dec 1;26(34):5504-10. doi: 10.1200/JCO.2008.17.9788. Epub 2008 Oct 27. PMID 18955447
- [Background] Jimeno A, Chan A, Cusatis G, Zhang X, Wheelhouse J, Solomon A, Chan F, Zhao M, Cosenza SC, Ramana Reddy MV, Rudek MA, Kulesza P, Donehower RC, Reddy EP, Hidalgo M. Evaluation of the novel mitotic modulator ON 01910.Na in pancreatic cancer and preclinical development of an ex vivo predictive assay. Oncogene. 2009 Jan 29;28(4):610-8. doi: 10.1038/onc.2008.424. Epub 2008 Nov 24. PMID 19029951
- [Background] Reddy MV, Mallireddigari MR, Cosenza SC, Pallela VR, Iqbal NM, Robell KA, Kang AD, Reddy EP. Design, synthesis, and biological evaluation of (E)-styrylbenzylsulfones as novel anticancer agents. J Med Chem. 2008 Jan 10;51(1):86-100. doi: 10.1021/jm701077b. Epub 2007 Dec 19. PMID 18088089
- [Background] Gumireddy K, Reddy MV, Cosenza SC, Boominathan R, Baker SJ, Papathi N, Jiang J, Holland J, Reddy EP. ON01910, a non-ATP-competitive small molecule inhibitor of Plk1, is a potent anticancer agent. Cancer Cell. 2005 Mar;7(3):275-86. doi: 10.1016/j.ccr.2005.02.009. PMID 15766665
- [Result] Garcia-Manero G, Fenaux P. Comprehensive Analysis of Safety: Rigosertib in 557 Patients with Myelodysplastic Syndromes (MDS) and Acute Myeloid Leukemia (AML). Blood Dec 2016, 128 (22) 2011; ASH 2016.
- See also: Website of St. Vincent Health, one of the clinical sites conducting the study. Information about St. Vincent Health, links to other related sites. — http://www.stvincent.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at one site in the United States. One patient was enrolled and treated, after which, the study was closed due to slow enrollment.
Period: Overall Study
Arm/Group | ON 01910.Na
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | ON 01910.Na
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: Progression-free survival, defined as the number of days from the first day of study drug dosing to the day of documented disease progression or death, as assessed using RECIST (Response Evaluation Criteria in Solid Tumors) guidelines according to Therasse P, Arbuck SF, Eisenhauer EA, et al. (2000) J Natl Cancer Inst. 92:205-216. Progressive disease is defined as at least a 20% increase in the sum of the longest diameter (LD)of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: 6 months
Measure: Number; unit: day
Arm/Group | ON 01910.Na
Number analyzed (Participants) | 1
day | 54

2. Secondary Outcome: Number of Adverse Events
Description: The number of adverse events and their severity rating will be classified according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events, version 3.0.
Time Frame: 6 months
Measure: Number; unit: Adverse event
Arm/Group | ON 01910.Na
Number analyzed (Participants) | 1
Adverse event | 9

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | ON 01910.Na
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ON 01910.Na (N=1)
Hypomagnesia (Metabolism and nutrition disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Pain-right flank (Musculoskeletal and connective tissue disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Investigators agree to inform the Sponsor of any publication or presentations on the study. All manuscripts, abstracts or presentations (in outline form with copies of slides if available) will be submitted to the Sponsor at least 30 days prior to the submission of the data for publication in order for the Sponsor to protect proprietary information. The Sponsor will review the submitted material within a reasonable period of time and will not unreasonably withhold publication permission.